CLINICAL TRIAL: NCT06445998
Title: Effect of Task Oriented Training on Cognitive Function in Elderly Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Horus University (Other)
Responsible Party: Principal Investigator, Ahmed Metwally Mohamed Elshinnawy, Assistant Professor, Department of Physical Therapy for Neuromuscular Disorders and Its Surgery, Faculty of Physical Therapy, Horus University, New Damietta, Egypt, Horus University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HorusU
Record Dates: First submitted 2024-06-01; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Stroke
Keywords: Task Oriented Training - Cognitive Function
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: task oriented training
Who Masked: Participant
Masking Description: traditional physical therapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (study group) (Experimental): consisted of twenty hemiparetic patients received task oriented training in addition to traditional physical therapy program, 3 times per week for 3 month, every session for 1 hour (30 minutes task oriented training followed by 30 minutes traditional physical therapy program).
  Interventions: Other: task oriented training
- Group B (control group) (Active Comparator): consisted of twenty hemiparetic patients received the traditional physical therapy program, 3 sessions/week for 3 month, each session for 1hour.
  Interventions: Other: task oriented training

INTERVENTIONS:
Other: task oriented training — Task-oriented training program: [For study group] Rocker board training Wobble board training Sit to stand Walk five steps forward Upstairs and downstairs three steps

SUMMARY:
Background: The impact of stroke at the time of diagnosis is on the attention and executive functions, which may be impaired at various post-stroke intervals. Objective: To improve Cognitive Function in Elderly Stroke Patients through Task Oriented Training. Subjects and methods: Forty Elderly stroke patients from both sexes assigned randomly into two equal groups. In Group A were allocated to task oriented training in addition to traditional physical therapy program, group B received traditional physical therapy program, three sessions/week for 3 months. Cognitive Function assessed by Reha-com device, Addenbrooke's Cognitive Examination Revised (ACE-R) test and Montreal Cognitive Assessment Scale (MoCA), measured at baseline and after 3 months.

DETAILED DESCRIPTION:
Methods The current study was conducted to examine the influence of task oriented training on cognitive functions in post Elderly stroke patients. All patients were diagnosed clinically and radiologically and referred from their neurological consultants as having post stroke cognitive impairment (PSCI). The patients were chosen, and the study was carried- out in outpatient clinics of Faculty of physical therapy, Horus University, this study was conducted at the period from ============== to==============.

True experimental research design study (one factorial RCT, pre-test and post-test control group design) was utilized. One trained research assistant assessed all patients and collected all data to reduce inter-investigator error. Patients were randomized according to the treatment procedure into two equal groups.

Randomization method: Patients who met the study's inclusion criteria were randomized into two groups (A and B) utilizing a secure opaque closed envelope allocation mechanism. Group A (study group): consisted of twenty hemiparetic patients received task oriented training in addition to traditional physical therapy program, 3 times per week for 3 month, every session for 1 hour (30 minutes task oriented training followed by 30 minutes traditional physical therapy program). Group B (control group): consisted of twenty hemiparetic patients received the traditional physical therapy program, 3 sessions/week for 3 month, each session for 1hour.

Blinding: All patients were assessed and referred by the same physician and physical therapy evaluation before beginning and at the end of the treatment program. Treatment allocations were kept secret from both the researcher and the participants.

Inclusion criteria: Forty right-handed hemiparetic patients from both genders aged from 60 to 70 years old. They are complaining from a single ischemic stroke diagnosed by Neurologist and confirmed radiologically by MRI of the brain. Duration of illness ranged from three to twelve months. Spasticity grade (1 to 1+) based on the Modified Ashworth Scale (MAS). Medically as well as psychologically stable patients. All patients had normal and stable vital signs (heart rate, blood pressure, temperature as well as respiratory rate). All patients had a good educational level and the body mass index ranged from 20-30 Kg/m2.

Exclusion criteria: Patients with Recurrent stroke or hemiparesis due to other neurological causes rather than stroke. Patients with severe cardiovascular issues that have not been adequately treated. Visual, auditory and other neurological disorders. Patients receiving medications that may affect cognition.

Data collection and intervention Assessment methods After being informed of the study's goals, methods, potential benefits, privacy, as well as data use, all participants signed a written consent form. Pre-treatment and post-treatment assessments were conducted on all patients.

Measurement procedures:

1. Assessment of cognitive function by Reha-com device The computerized Reha-Com device containing the (attention and concentration) program was utilized as the patient is asked to concentrate on every detail in the separately presented picture and select the one that resembles it in every detail from the matrix, as the assessment screen is splitted into two parts. One portion represents the matrix that involves: according to (24) levels of difficulty: 3 pictures (1 by 3 matrix), 6 pictures (2 by 3 matrix) as well as 9 pictures (3 by 3 matrix), and the other part represents the separated picture.
2. Addenbrooke's Cognitive Examination Revised (ACE-R) test It consists of 26 tasks, divided into five domains. It takes about 15 minutes to administer. The maximum possible score is 100, and questions are asked in the sequence stated, with scores calculated immediately based on the addition of point values for each correctly answered question (10).
3. Montreal Cognitive Assessment Scale (MoCA):

The test is commonly used to screen for cognitive impairment. It was designed to detect mild cognitive Impairment. It takes approximately 10 minutes to complete, 30-point cognitive screening instrument. It is utilized to evaluate multiple aspects of cognition, including: short-term memory; visual-spatial skills; executive function; concentration; attention; memory for work; language; as well as time-and-place awareness. The possible range of MoCA scores is 0-30. If you scored 26 or more, you're in the normal range. Scores below 25 indicate mild cognitive impairment (MCI) in individuals who have suffered a stroke, and the score has a high sensitivity (77%) as well as specificity (83%) (11).

Intervention methods Task-oriented training program: [For study group] Rocker board training The subject was asked to control anteroposterior then mediolateral rolling movement of the rocking board, first placing both feet then one foot, first with eyes opened then with eyes closed, from sitting then standing position.

Wobble board training The subject was asked to try to stop the multidirectional rolling wobble board movement, first with eyes opened then with eyes closed, from sitting then standing position, repeat 10 times.

Sit to stand The patient was instructed to lean forward then press on heel then stand up. Both hands should be on the thigh and push against it to stand. This progress to be performed with opened eyes then with closed eyes firstly on a firm surface then on foam surface with repetitions 10 times.

Walk five steps forward From standing position, the patient was asked to walk five steps forward firstly on a firm surface, then on foam surface and repeat 10 times.

Upstairs and downstairs three steps The patient was asked to perform upstairs five steps and downstairs with hand supported then without hand supported, repeat 10 times.

Traditional physical therapy program: [For both groups] Range of motion exercises Range of motion exercises was performed for the foot. The patient was asked to sit in a chair, lift the affected foot and circle in a clockwise, then a counterclockwise motion. Repeat this cycling five and ten times in each direction.

Strengthing exercises:

Graduate active exercise was used through strengthing of ankle dorsiflexors, planterflexor, invertors and evertors. Proprioceptive neuromuscular facilitation was also applied to strength distal muscles in the form of repeated contraction for dorsiflexors of ankle joint for ten minutes.

Sensory re-education:

Tactile stimulation for both superficial and deep sensation was applied. Gait Training Walking within parallel bar with hand supported then without hand support was participated for ten minutes. Obstacles also were used with hand support then without hand support.

ELIGIBILITY:
Inclusion criteria:

* Forty right-handed hemiparetic patients from both genders aged from 60 to 70 years old.
* They are complaining from a single ischemic stroke diagnosed by Neurologist and confirmed radiologically by MRI of the brain. Duration of illness ranged from three to twelve months. Spasticity grade (1 to 1+) based on the Modified Ashworth Scale (MAS).
* Medically as well as psychologically stable patients. All patients had normal and stable vital signs (heart rate, blood pressure, temperature as well as respiratory rate).
* All patients had a good educational level and the body mass index ranged from 20-30 Kg/m2.

Exclusion criteria:

* Patients with Recurrent stroke or hemiparesis due to other neurological causes rather than stroke.
* Patients with severe cardiovascular issues that have not been adequately treated. Visual, auditory and other neurological disorders.
* Patients receiving medications that may affect cognition.

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
1- Assessment of cognitive function by Reha-com device | 3 month
  The computerized Reha-Com device containing the (attention and concentration) program was utilized as the patient is asked to concentrate on every detail in the separately presented picture and select the one that resembles it in every detail from the matrix, as the assessment screen is splitted into two parts. One portion represents the matrix that involves: according to (24) levels of difficulty: 3 pictures (1 by 3 matrix), 6 pictures (2 by 3 matrix) as well as 9 pictures (3 by 3 matrix), and the other part represents the separated picture.
2- Addenbrooke's Cognitive Examination Revised (ACE-R) test | 3 month
  It consists of 26 tasks, divided into five domains. It takes about 15 minutes to administer. The maximum possible score is 100, and questions are asked in the sequence stated, with scores calculated immediately based on the addition of point values for each correctly answered question (10).
3- Montreal Cognitive Assessment Scale (MoCA): | 3 month
  The test is commonly used to screen for cognitive impairment. It was designed to detect mild cognitive Impairment. It takes approximately 10 minutes to complete, 30-point cognitive screening instrument. It is utilized to evaluate multiple aspects of cognition, including: short-term memory; visual-spatial skills; executive function; concentration; attention; memory for work; language; as well as time-and-place awareness. The possible range of MoCA scores is 0-30. If you scored 26 or more, you're in the normal range. Scores below 25 indicate mild cognitive impairment (MCI) in individuals who have suffered a stroke, and the score has a high sensitivity (77%) as well as specificity (83%) (11).

CONTACTS AND LOCATIONS:
Overall Officials: Zeezy S Eraky, Lecturer, Study Chair — Department of Physical Therapy for Internal Medicine and Elderly; Haitham M. Elmasry, Lecturer, Study Chair — Department of Basic Science; Ibrahim M. Hamoda, Asst Prof, Study Chair — Department of Physical Therapy for Neuromuscular Disorders and its Surgery
Locations (1):
- Horus University, Damietta, New Damietta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
All the IPD will be shared Through the Corresponding author after acceptance of all authors